CLINICAL TRIAL: NCT01372709
Title: A Post-Market Study to Evaluate the Safety and Performance of the Ovation™ or Ovation Prime™ Abdominal Stent Graft System
Brief Title: TriVascular Post-Market Registry
Status: Completed | Type: Observational
Sponsor: TriVascular, Inc. (Industry)
Responsible Party: Sponsor
Organization: Endologix (Industry)
Other Study IDs: 771-0008
Record Dates: First submitted 2011-06-10; First posted 2011-06-14 (Estimated); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: abdominal; aortic; aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ovation™ or Ovation Prime™ Abdominal Stent Graft System: Adult male and female patients will be consecutively screened for the study. Eligible patients must meet all of the inclusion criteria and none of the exclusion criteria.
  Interventions: Device: Ovation™ or Ovation Prime™ Abdominal Stent Graft System

INTERVENTIONS:
Device: Ovation™ or Ovation Prime™ Abdominal Stent Graft System — Single occurrence permanent implant of AAA device.

SUMMARY:
This is a prospective observational post-market study of subjects receiving the Ovation™ or Ovation Prime™ Abdominal Stent Graft System ("Ovation™ or Ovation Prime™ Abdominal Stent Graft System Post-Market Study") in the treatment of abdominal aortic aneurysms (AAA). The Ovation™ or Ovation Prime™ Abdominal Stent Graft System Post-Market study is intended to expand the clinical knowledge base by collecting data on subjects treated with the Ovation™ or Ovation Prime™ Abdominal Stent Graft System in actual clinical practice following commercial approval.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years or minimum age as required by local regulations.
* Indication for elective repair of AAA with an endovascular stent graft in accordance with the Instructions for Use of the Ovation™ or Ovation Prime™ Abdominal Stent Graft System.
* Subject has signed an Ethics Committee (EC) approved Informed Consent Form. The subject or legal representative has been informed of the nature of the study, has consented to participate, and has authorized the collection and release of his/her medical information.
* Subject intends to electively receive the Ovation™ or Ovation Prime™ Abdominal Stent Graft System.
* Subject has the ability and willingness to comply with all follow-up exams as indicated in clinical investigation plan.

Exclusion Criteria:

* Subject demonstrates high probability of non-adherence to physician's follow-up requirements.
* Subject's current participation in a concurrent randomized control trial (RCT) or investigational device/drug study which could confound study results.
* Life expectancy less than 1 year
* Pregnancy
* Subjects with poor renal function as indicated by a serum creatinine > 2.5mg/dl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Ovation™ or Ovation Prime™ Abdominal Stent Graft System study is a multicenter, prospective, observational post-market study of subjects receiving the Ovation™ or Ovation Prime™ Abdominal Stent Graft System for the treatment of abdominal aortic aneurysms (AAA). The Ovation™ or Ovation Prime™ Abdominal Stent Graft System Post-Market Study intends to expand the clinical evidence of the safety and performance of the Ovation™ or Ovation Prime™ Abdominal Stent Graft System in an all comers ("real world") patient population.
Sampling Method: Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2014-12-12 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Treatment Success at 12 Months Post-Implantation/surgery. | 12 Months
  The primary endpoint is treatment success at 12 months post-implantation/surgery. Treatment success is defined as a composite technical endpoint composed of successful introduction and deployment of the Ovation™ or Ovation Prime™ Abdominal Stent Graft System at the initial implantation procedure along with clinical endpoints of absence from type I or III endoleaks, aneurysm expansion, aneurysm rupture, conversion to open surgical repair, graft migration, and graft occlusion at 12 months post-implantation procedure.

SECONDARY OUTCOMES:
Safety and Performance Endpoints | 1, 6, &12 Months
  * Freedom from type I and III endoleaks [1 & 6 m, & annual through 5 years]
  * Freedom from aneurysm rupture [6 m, & annual through 5 years]
  * Freedom from aneurysm related mortality [1 month]
  * Freedom from aneurysm expansion [6 m, & annual through 5 years]
  * Freedom from stent graft migration [6 m, & annual through 5 years]
  * Freedom from loss of device patency [1 & 6 m, & annual through 5 years]
  * Freedom from aneurysm-related secondary endovascular procedures [1 & 6 m, & annual through 5 years]
  * Freedom from device related adverse events [1 & 6 m, & annual through 5 years]

CONTACTS AND LOCATIONS:
Locations (30):
- Medical University of Vienna Dept. for Radiology, Section for Cardiovascular and Interventional Radiology, Vienna, Austria
- Belgium (5):
  - O.L. Vrouwziekenhuis, Aalst
  - Imelda Ziekenhuis, Bonheiden
  - Flanders Medical Research Program, Dendermonde
  - Universiteit Gent, Ghent
  - UZ Leuven, Leuven
- France (2):
  - Groupe Hospitalier Edouard Herriot, Lyon
  - Hôpital Paul d'Egine, Paris
- Germany (7):
  - Park Hospital Leipzig, Strümpellstr. 41, Leipzig, Western Saxony Land
  - Herz- und Gefässzentrum Bad Bevensen, Bad Bevensen
  - Franziskus-Krankenhaus Berlin, Berlin
  - Cardiovascular Center, Frankfurt
  - Universitäres Herz und Gefaßzentrum Hamburg, Hamburg
  - Städtisches klinikum Karlsruhe Klinik für Gefäß- und Thoraxchirurgie, Karlsruhe
  - "CA Gefäßchirurgie Theresienkrankenhaus/St. Hedwig", Mannheim
- Attikon Hospital, Athens, Greece
- Italy (10):
  - Ospedale San Raffaele, Milan
  - Policlinico San Donato, Milan
  - Ospedale Civico Palermo, Palermo
  - Ospedale Bianchi Melacrino Morelli, Reggio Calabria
  - Azienda Ospedaliera Sant'Andrea, Roma
  - Ospedale San Giovanni Addolorata, Roma
  - Università La Sapienza/Policlinico Umberto I, Roma
  - Univeristà La Sapienza/Policlinico Umberto I, Rome
  - Ospedale San Giovanni Bosco, Torino
  - A.O. Ospedale di Circolo e Fondazione Macchi, Varese
- Södersjukhuset, Stockholm, Sweden
- United Kingdom (3):
  - Frimley Park Hospital NHS Foundation Trust, Frimley
  - St. George's Vascular Institute, London
  - Manchester Royal Infirmary, Manchester